CLINICAL TRIAL: NCT00308555
Title: Opioid and Cannabinoid Pharmacokinetic Interactions: A Pilot Study
Brief Title: Opioid and Cannabinoid Pharmacokinetic Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC # 064; 1R21DA020831-01 (NIH)
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: Cannabis; Morphine; Oxycodone; Marijuana; chronic pain
MeSH Terms: conditions — Pain; Marijuana Abuse; Chronic Pain | interventions — nabiximols

ARMS (1):
- Cannabis (Other)
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis

SUMMARY:
We are conducting a study to assess whether smoking marijuana affects the safety of prescribed opioids in patients treated for chronic pain. This study will assess whether smoking cannabis affects the absorption, distribution, metabolism and excretion of widely used opioid analgesics. We propose to do this by investigating the effects of smoked cannabis in subjects prescribed morphine or oxycodone for chronic pain. We will also assess the clinical safety of cannabinoids and these opioids by monitoring the short-term side effects associated with combined therapy.

DETAILED DESCRIPTION:
Chronic pain conditions remain problematic, especially in patients with cancer. Although opioids are effective analgesics, dose-limiting side effects in the form of sedation, nausea and vomiting, and fear of dependence often limit their use at higher - and possibly more effective - doses. Of particular interest, however, is the potential for greater than additive analgesic effect of cannabinoids and opioids in combination that would allow for opioid analgesic effect to be achieved at lower dosages than are necessary alone, which could overcome problems with both tolerance and side effects for both drug classes. Unfortunately, safety data on the combination in humans does not exist at this time and needs to be obtained. As increasing numbers of patients with chronic pain may turn to cannabis to augment the effects of their opioid analgesics, data on potential pharmacokinetic interactions and clinical safety of the combinations should be evaluated in a controlled clinical research setting.

ELIGIBILITY:
Inclusion Criteria:

1. Ongoing analgesic therapy with either oxycodone hydrochloride (OxyContin) or morphine sulfate (MS Contin) every 12 hours for chronic pain.
2. Eligible subjects will be ≥ 18 years of age with a diagnosis of chronic pain and an estimated survival of greater than six months.
3. Subjects must be on a stable dose of opioid medication for at least 2 weeks before enrollment.
4. Current other analgesic medications will be maintained during the study. The subject must have been on a stable medication regimen for at least 2 weeks.
5. The following laboratory parameters documented within 45 days prior to study entry:

   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 X upper limit of normal (ULN)
   * Total bilirubin ≤ 2 X ULN
   * Creatinine ≤ 2.0 mg/dL (177 µmol/L)
6. All men and women in this study must agree to use adequate birth control during this study. Acceptable barrier birth control methods are a male condom, female condom, diaphragm, or intra-uterine (IUD).
7. All women of reproductive potential (who have not reached menopause or undergone hysterectomy, oophorectomy, or tubal ligation) must have a negative urine b-HCG pregnancy test performed before initiating the protocol-specified medication.
8. Prior history of use of marijuana. Subjects must have smoked marijuana on at least 6 occasions in their lifetime prior to enrollment.
9. Able to understand and follow the instructions of the investigator, including completing the pain intensity rating scales.
10. Karnofsky Performance Score >60.
11. Able and willing to provide informed consent.

Exclusion Criteria:

1. Severe coronary artery disease, uncontrolled hypertension, cardiac ventricular conduction abnormalities, or orthostatic mean blood pressure drop greater than 24 mmHg, severe chronic obstructive pulmonary disease.
2. History of renal or hepatic failure.
3. Evidence of hepatic, hematological or renal dysfunction based on judgment of physician.
4. Active substance abuse (e.g., alcohol or injection drugs).
5. Use of smoked marijuana within 30 days of enrollment verified with a urine THC level.
6. Neurologic dysfunction or psychiatric disorder severe enough to interfere with assessment of pain or sensory systems.
7. Current use of smoked tobacco products or a confirmed cotinine level.
8. Women who are pregnant or breast-feeding may not take part in this study.
9. Unable to read or speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald I Abrams, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Community Consortium, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 315 participants were screened, via phone and e-mail, between January 2007 and February 2009. 24 subjects were enrolled, 13 taking morphine and 11 taking oxycodone.
Groups:
- MS Contin: Patients using morphine sulfate (MS Contin) every 12 hours for chronic pain were administered vaporized cannabis (3.96% delta 9-THC) equivalent to one 0.9 g cigarette on the following schedule: 20:00 on Day 1, 08:00/14:00/20:00 on Days 2 through 4, and 08:00 on Day 5.
- Oxycontin: Patients using oxycodone hydrochloride (OxyContin) every 12 hours for chronic pain were administered vaporized cannabis (3.96% delta 9-THC) equivalent to one 0.9 g cigarette on the following schedule: 20:00 on Day 1, 08:00/14:00/20:00 on Days 2 through 4, and 08:00 on Day 5.
Period: Overall Study
Arm/Group | MS Contin | Oxycontin
Started | 13 | 11
Completed | 10 | 11
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- MS Contin: Patients using morphine sulfate (MS Contin) every 12 hours for chronic pain
- Oxycontin: Patients using oxycodone hydrochloride (OxyContin)every 12 hours for chronic pain
- Total: Total of all reporting groups
Arm/Group | MS Contin | Oxycontin | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (7.4) | 47.1 (11.8) | 45.1 (10.0)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24
Mean opioid dose, twice daily [Mean (Full Range); unit: mg] — Baseline medication use
  mg | 62 [10 to 100] | 53 [10 to 120] | 58 [10 to 120]

OUTCOME MEASURES:

1. Primary Outcome: Disposition Kinetics of Morphine and Oxycodone Before and After Cannabis Use
Description: Pharmacokinetics are measured on Day 1, prior to cannabis use, and again on Day 5, following cannabis use on Days 2, 3, and 4.
Time Frame: Day 1, Day 5
Population: The number was determined by the number of participants completing both Day 1 and Day 5 procedures.
Measure: Number (95% Confidence Interval); unit: Geometric Mean Ratio
Groups:
- MS Contin: Participants on morphine treatment
- Oxycodone: Participants on oxycodone treatment
Arm/Group | MS Contin | Oxycodone
Number analyzed (Participants) | 10 | 11
Geometric Mean Ratio
  Time to maximum concentration (Tmax) | 1.64 [-1.01 to 4.30] | -1.11 [-3.66 to 1.43]
  Maximum concentration (Cmax) | 0.9 [0.85 to 0.95] | 0.99 [0.89 to 1.10]
  Area under plasma concentration-time curve (AUC) | 0.95 [0.84 to 1.05] | 0.94 [0.84 to 1.04]

ADVERSE EVENTS:
Groups:
- MS Contin: Patients using morphine sulfate (MS Contin) every 12 hours for cancer pain
- Oxycontin: Patients using oxycodone hydrochloride (OxyContin)every 12 hours for cancer pain
Arm/Group | MS Contin | Oxycontin
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

LIMITATIONS AND CAVEATS:
Small number of participants, powered to detect a 25% change in AUC(12).Further research is needed to determine how cannabis delivery systems other than vapor affect metabolism of opioids and other drugs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No